CLINICAL TRIAL: NCT05087667
Title: Outcomes of Adjuvant "Polymer Cerclage System "OrthoLoop" to Manage Prosthetic Rehabilitation, Per Prosthetic or Primary Femoral and Humeral Fractures. a Prospective , Multicentric, Simple Blind , Comparative, Non-inferiority Study, Compared to Cerclage Systems Used in Standard Care.
Brief Title: Study of the Effectiveness of a Polymer Cerclage System Compared to Cerclages Used in Standard Care (CERCPMCF) )
Acronym: SERRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quanta Medical (Industry)
Collaborators: Cousin Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3069_CERCPMCF
Record Dates: First submitted 2021-09-21; First posted 2021-10-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-11

CONDITIONS: Femoral Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Intervention Model Description: Cluster's randomization
Who Masked: Participant
Masking Description: Single blinded study. The patient will be blinded from the randomization arm. As the procedure is performed under general anaesthesia, the patient will not be informed whether or not the Sterile Self Locking Polymer Cerclage System has been implanted as a result of the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polymer Cerclage System OrthoLoop (Experimental): Patients receives Ortholoop Cerclage System
  Interventions: Device: Implantation of Ortholoop cerclage
- cerclages used in standard care (Active Comparator): Patients receives cerclages used in standard care"
  Interventions: Device: Implantation of Cerclage used in current practice

INTERVENTIONS:
Device: Implantation of Ortholoop cerclage — implantation of Sterile Self Locking Polymer Cerclage System named OrthoLoop to the patient and follow up for 36 months post-intervention
  Arms: Polymer Cerclage System OrthoLoop
Device: Implantation of Cerclage used in current practice — implantation of Cerclage used in current practice to patients and follow up for 36 months post-intervention
  Arms: cerclages used in standard care

SUMMARY:
The use of cerclage wiring in the management of long bone fractures is common. With the increase in the placement of total hip ans shoulder prostheses, the occurrence of peri-prosthetic hip an shoulder fractures is also increasing, notably due to an older population.

Whether it is for a fracture on a native femur or humerus, or on a periprosthetic hip or shoulder fracture, the use of cerclage wiring is an adjuvant additional but not the main means to ensure stable osteosynthesis, allowing re-loading and early rehabilitation of patients. This method has demonstrated its ability to improve the fixation of this fracture type, associated with osteosynthesis or hip/shoulder prosthesis revision surgery. However, metal cerclage expose to a risk of metallosis which can compromise bone fusion, injury to neighboring soft parts causing pain and also injury to the surgical team when handling them. More recently, non-metallic cerclage have been developed and could overcome certain risks associated with metallic cerclage, while ensuring their bone fixing capacity and therefore bone consolidation. Indeed, non-metallic cerclage could withstand similar or even greater stresses than metallic cables, in particular concerning their resistance to rupture.

The "Sterile Self Locking Polymer Cerclage System" named OrthoLoop is a polymer cerclage which has been developed and could be used in these indications.

Thus, this study (SERRE) aims to investigate the clinical results and sequelae of adjuvant cerclage wires OrthoLoop Cerclage in the management of rehabilitation, per prosthetic or primary femoral or humeral fractures compared with cerclages system used in standard care.

SERRE is a 36 months follow up study in two arms :

* Experimental group: "OrthoLoop cercalge"
* Control group: "cerclages used in standard care" After each surgery, the patient follow-up period is 36 months. with 4 planned consultation visits after surgery at 6-8 weeks, 3, 6 and 36 months, with collection and measurement of the endpoints.

The main objective of this study is to assess the role of "OrthoLoop cerclage" of COUSIN Biotech in comparison with cerclages (metallic for the majority) used in standard care ; in the optimization of the consolidation of primary and periprosthetic femoral or humeral fractures, 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient with femoral or humeral fracture requiring the installation of one or more cerclage(s) and respecting at least one of the criteria below:
* Primary femoral or humeral fractures (diaphyseal, metaphyseal, epiphyseal proximal or distal) with osteosynthesis by plate and screw or osteosynthesis by Intramedullary nailing associated with the installation of one or more cerclage(s)
* Patients with traumatic fracture of femur or humerus that required prosthetic rehabilitation associated with the installation of one or more cerclage(s)
* Peri-prosthetic fracture of the femur or humerus
* Resumption of prosthesis (hip, knee, shoulder, elbow) requiring the installation of one or more cerclages
* who underwent fixation with cerclage wiring (Sterile Self Locking Polymer Cerclage System or other cerclage systems used in standard care)
* age ≥18 years
* Who have given free, informed and written consent to participate in the study
* Patient able to communicate in French
* Patient affiliated to a social security system or entitled to a social security system

Exclusion Criteria:

* high-energy injury,
* associated damage to other long bones,
* fracture extension to the articular surface with displacement
* Severe disease that could interfere with the study results or be life threatening
* Patients with an infection
* Allergy to any component of the medical products
* Pregnant or breastfeeding women
* Anticipated unavailability during the study
* Participation in a clinical trial within 3 months prior to the inclusion visit.
* Patient with linguistic or psychological incapacity to understand and sign the informed consent.
* Patient deprived of liberty by administrative or judicial decision, or being under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Assess role of Polymer Cerclage System OrthoLoop of COUSIN Biotech in comparison with cerclages (metallic for the majority) used in standard care; in the optimization of the consolidation of primary and periprosthetic fractures of long bones | 6 months post-surgery
  primary endpoint will be success or failure 6 months after surgery:
  Success of "Sterile Self Locking Polymer Cerclage System" to optimize consolidation during 6 months post surgery is defined as:
  * the ability to walk full weight bearing without pain at the fracture site, or return to normal, painless mobility at the fracture site,
  * and radiographs showing signs of bony union with no rupture or migration of the cerclage.
  Rupture or cerclage migration or nonunion or need for revision of the implant before 6 months is considered as failure.

SECONDARY OUTCOMES:
Assess consolidation rate during 6 months post surgery | 6 months post-surgery
  Consolidation (or union) is defined as the ability to walk full weight bearing without pain or return to normal, painless mobility at the fracture site , and radiographs showing signs of bony union
Asses union time | 3, 6 and 36 months post-surgery
  Union time is defined as time from intervention until
  * For Femoral fracture: ability of patient to walk full weight bearing without pain at the fracture site and radiographs showing signs of bony union
  * For humeral fracture: The patient regained full mobility without pain at the fracture site.
Assess rupture and migration rate of the cerclage after surgery throughout the follow-up | 3, 6 and 36 months post-surgery
  Rupture and migration of the cerclage are confirmed on X Ray imaging.
Assess pain | 6-8 weeks,3, 6 and 36 months post-surgery
  Pain will be assessed using visual analog scale pain scores (VAS) from 0 to 100 (0 means no pain at all and 100 maximum pain) at each visit.
To report the incidence of complications and their treatment, particularly with respect to the need of further surgery | During the whole study (up to 36 months)]
  Safety data during patients 36 months follow up are defined such as:
  Infection Neurovascular injury Allergic reaction Bone ischemia Irritation feeling
Assess surgery characteristics | During surgery (at D0)
  Surgery characteristics are:
  Rupture of cerclage during the surgery (at time of implantation) Number of wire cerclages used implant used for osteosynthesis (nail or plate) Using of screw fixation operative time
Assess physicians satisfaction regarding the use of "Sterile Self Locking Polymer Cerclage System | During surgery (at D0)
  Physicians satisfaction regarding the use of "Sterile Self Locking Polymer Cerclage System" will be assessed on:
  Global satisfaction of the surgeon Ease of use Ancillaries (Cable Passer, Tensioner) : ease of use and lightweight Ease of tension control by the surgeon using tensioner Ease of tracking of the cerclage on radiography Resistance over time (at least until bone consolidation) Presentation (ease of unwinding, packaging)

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - Clinique ESQUIROL SAINT HILAIRE, Agen, France
  - Hôpital Privé Francheville, Périgueux, France
  - CH Tourcoing, Tourcoing, France
  - CHU Lille, Lille, Nord
  - CH Agen, Agen
  - CH Arcachon, Arcachon
  - Clinique de Saint Omer, Blendecques
  - CH Le Mans, Le Mans
  - CH Libourne, Libourne
  - Ch Metz - Thionville, Metz
  - CHRU Nancy, Nancy
  - CHU Nimes, Nîmes
  - Polyclinique Du Parc, Saint-Saulve
  - CHU Toulouse, Toulouse
  - CH Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindahl H. Epidemiology of periprosthetic femur fracture around a total hip arthroplasty. Injury. 2007 Jun;38(6):651-4. doi: 10.1016/j.injury.2007.02.048. Epub 2007 May 2. PMID 17477925
- [Background] Rayan F, Haddad F. Periprosthetic femoral fractures in total hip arthroplasty - a review. Hip Int. 2010 Oct-Dec;20(4):418-26. doi: 10.1177/112070001002000402. PMID 21157744
- [Background] Tsiridis E, Pavlou G, Venkatesh R, Bobak P, Gie G. Periprosthetic femoral fractures around hip arthroplasty: current concepts in their management. Hip Int. 2009 Apr-Jun;19(2):75-86. doi: 10.1177/112070000901900201. PMID 19462362
- [Background] Ferbert T, Jaber A, Gress N, Schmidmaier G, Gotterbarm T, Merle C. Impact of intraoperative femoral fractures in primary hip arthroplasty: a comparative study with a mid-term follow-up. Hip Int. 2020 Sep;30(5):544-551. doi: 10.1177/1120700019849911. Epub 2019 May 17. PMID 31096789
- [Background] Ebraheim NA, Sochacki KR, Liu X, Hirschfeld AG, Liu J. Locking plate fixation of periprosthetic femur fractures with and without cerclage wires. Orthop Surg. 2013 Aug;5(3):183-7. doi: 10.1111/os.12052. PMID 24002835
- [Background] Angelini A, Battiato C. Combination of low-contact cerclage wiring and osteosynthesis in the treatment of femoral fractures. Eur J Orthop Surg Traumatol. 2016 May;26(4):397-406. doi: 10.1007/s00590-016-1761-3. Epub 2016 Mar 17. PMID 26983607
- [Background] Gordon K, Winkler M, Hofstadter T, Dorn U, Augat P. Managing Vancouver B1 fractures by cerclage system compared to locking plate fixation - a biomechanical study. Injury. 2016 Jun;47 Suppl 2:S51-7. doi: 10.1016/S0020-1383(16)47009-9. PMID 27338228
- [Background] Angelini A, Battiato C. Past and present of the use of cerclage wires in orthopedics. Eur J Orthop Surg Traumatol. 2015 May;25(4):623-35. doi: 10.1007/s00590-014-1520-2. Epub 2014 Sep 4. PMID 25186972
- [Background] Altenburg AJ, Callaghan JJ, Yehyawi TM, Pedersen DR, Liu SS, Leinen JA, Dahl KA, Goetz DD, Brown TD, Johnston RC. Cemented total hip replacement cable debris and acetabular construct durability. J Bone Joint Surg Am. 2009 Jul;91(7):1664-70. doi: 10.2106/JBJS.G.00428. PMID 19571089
- [Background] Silverton CD, Jacobs JJ, Rosenberg AG, Kull L, Conley A, Galante JO. Complications of a cable grip system. J Arthroplasty. 1996 Jun;11(4):400-4. doi: 10.1016/s0883-5403(96)80029-5. PMID 8792246
- [Background] Peeters I, Depover A, Van Tongel A, De Wilde L. A review of metallic and non-metallic cerclage in orthopaedic surgery: Is there still a place for metallic cerclage? Injury. 2019 Oct;50(10):1627-1633. doi: 10.1016/j.injury.2019.06.034. Epub 2019 Jul 13. PMID 31326103